CLINICAL TRIAL: NCT04283227
Title: An Open Label, Non-randomized Trial to Evaluate the Safety and Efficacy of a Single Infusion of OTL-200 in Patients With Late Juvenile (LJ) Metachromatic Leukodystrophy (MLD).
Brief Title: OTL-200 in Patients With Late Juvenile Metachromatic Leukodystrophy (MLD)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Orchard Therapeutics (Industry)
Collaborators: Ospedale San Raffaele (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTL-200-07
Record Dates: First submitted 2020-02-13; First posted 2020-02-25 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Lysosomal Storage Diseases; Metachromatic Leukodystrophy
Keywords: OTL-200; Cryopreserved formulation; Gene therapy; MLD; late juvenile; atidarsagene autotemcel
MeSH Terms: conditions — Lysosomal Storage Diseases; Leukodystrophy, Metachromatic

STUDY DESIGN:
Intervention Model Description: All eligible subjects will receive intravenous (IV) infusion of OTL-200 gene therapy. Subjects will also receive conditioning regimen with busulfan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OTL-200 Gene Therapy (Experimental): OTL-200 is an autologous CD34+ cell enriched population that contains hematopoietic stem and progenitor cells (HSPC) transduced ex vivo using a lentiviral vector encoding the human arylsulfatase A (ARSA) gene.
  Interventions: Genetic: OTL-200

INTERVENTIONS:
Genetic: OTL-200 — All subjects will receive OTL-200 gene therapy and will be followed up for 8 years following treatment with OTL-200.

SUMMARY:
OTL-200 is a cryopreserved dispersion for infusion containing autologous CD34+ cell enriched population that contains haematopoietic stem and progenitor cells (HSPC) transduced ex vivo using a lentiviral vector encoding the human arylsulfatase A (ARSA) gene. MLD is an autosomal recessive lysosomal storage disorder (LSD) characterized by severe and progressive demyelination affecting the central and peripheral nervous system. The aim of this clinical study is to assess the pharmacodynamic effect and long-term clinical efficacy and safety of OTL-200 in Late Juvenile MLD patients.

ELIGIBILITY:
Inclusion Criteria:

All the following criteria need to be met:

* Documented biochemical and molecular diagnosis of MLD, based on ARSA activity below the normal range and identification of two disease-causing ARSA alleles. Novel mutations will be analyzed with in silico prediction tools and excluded from being known common polymorphisms. In the case of a novel mutation(s), a 24-hour urine collection must show elevated sulfatide levels.
* 0/R or R/R genotype or a genotype recognized as associated with the LJ variant of MLD.
* a) If symptomatic: age at disease onset between ≥7 and <17 years of age (i.e. before their 17th birthday). OR
* b) If pre-symptomatic: participant must be <17 years of age at treatment (i.e. before their 17th birthday) AND must have a sibling with a diagnosis of late-juvenile MLD variant based on age at disease onset (≥7 and <17 years of age i.e. before sibling's 17th birthday), with biochemical and molecular diagnosis.
* Normal cognitive function as defined by an IQ≥85 on age appropriate cognitive scales.
* a) If the participant is <7 years (i.e. before their 7th birthday): normal motor milestones achievement, normal gross motor function according to chronological age and normal neurological examination (if applicable based on the age of the subject, GMFC-MLD = 0) OR b) If participant is ≥7 years: normal gross motor function or mild gross motor function impairment, defined by a GMFC-MLD 0 or 1 (i.e. patient is able to walk independently).

NOTE: The following will not be exclusionary if present alone: 1.) Seizures 2.) Signs of the disease revealed at instrumental evaluations (Electroneurography [ENG] and brain MR)

* If applicable, participant willing and capable of compliance with contraceptive use requirements.
* Participant (or if applicable, parent/legal guardian) providing signed informed consent or assent as applicable

Exclusion Criteria:

* Documented HIV infection (positive HIV RNA and/or anti-p24 antibodies).
* Malignant neoplasia (except localised skin cancer) or a documented history of hereditary cancer syndrome. Participants with a prior successfully treated malignancy and a sufficient follow-up to exclude recurrence (based on oncologist opinion) can be included after discussion and approval by the Medical Monitor.
* Myelodysplasia, cytogenetic alterations characteristic of myelodysplastic syndrome (MDS) and acute myeloid leukaemia (AML) or other serious haematological disorders.
* Patients currently enrolled in other interventional trials
* Has previously undergone allogeneic HSPC gene therapy (HSPC-GT) and has evidence of residual cells of donor origin.
* Previous gene therapy.
* Has symptomatic herpes zoster, not responsive to specific treatment. NOTE: Participants with a recent history of herpes zoster may be included in the study. In such cases, inclusion, additional monitoring and treatment of the condition must be discussed and approved by the Medical Monitor.
* Evidence of active tuberculosis (TB) based upon medical examination, chest imaging and TB testing. Participants with latent tuberculosis, as documented by medical history and/or TB testing may be included in the study if receiving antibiotic prophylaxis (e.g. isoniazid). Inclusion, monitoring and treatment of TB in such participants must be discussed and approved by the Medical Monitor.
* Acute or chronic stable Hepatitis B (HBV) as evidenced by positive Hepatitis B surface antigen (HBsAg) test result at screening or within 3 months prior to onset of conditioning and/or positive HBV DNA. NOTE: Participants with positive Hepatitis B core antibody due to prior resolved disease may be enrolled, only if a confirmatory negative HBsAg and negative Hepatitis B DNA test are obtained. Inclusion, monitoring and treatment of hepatitis in such participants must be discussed and approved by the Medical Monitor.
* Presence of positive Hepatitis C RNA test result at screening. NOTE: Patients who have previously tested positive for antibodies to hepatitis C can be treated, provided they demonstrate absence of ongoing infection using a nucleic acid test with a limit of quantification of ≤15 international units/ml. Negative test results are required on at least 3 sequential occasions over a period of at least 4 weeks, after completion of treatment for Hepatitis C, with the final test conducted no more than 3 days prior to cell harvest. Inclusion, monitoring and treatment of hepatitis in such participants must be discussed and approved by the Medical Monitor.
* End-organ dysfunction, severe active infection not responsive to treatment, or other severe disease or clinical condition which, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* In addition to the potential infections tested per protocol, the PI should consider testing for other transmissible infectious agents listed in the European Union (EU) Cell and Tissue Directive as clinically appropriate and results must be discussed with the Orchard medical monitor prior to stem cell harvest.
* Participants with alanine transferase (ALT) >2x upper limit of normal (ULN) or total bilirubin >1.5xULN may be included only after discussed and agreed with the Orchard medical monitor and considered in the context of the criterion for excluding participants with other severe disease. Isolated elevation of total bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35% of total.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of OTL-200 Arylsulfatase A (ARSA) activity levels in Cerebrospinal Fluid (CSF) | 24 months after treatment
  Change from baseline in ARSA activity levels in CSF
Evaluation of OTL-200 on the neuronal metabolite ratio of N-acetyl-aspartate (NAA) to creatine (Cr) in white matter regions of the brain | 24 months after treatment
  Change from baseline in neuronal metabolite ratio of N-acetyl-aspartate (NAA) to creatine (Cr) in white matter regions of interest of the brain

SECONDARY OUTCOMES:
Change in ARSA activity levels in CSF from baseline | multiple visits up to 8 years post gene-therapy
  Measured to assess the pharmacodynamic activity of OTL-200 in the Central Nervous System (CNS) post-treatment
Change from baseline in neuronal metabolite ratio of NAA: Cr in white matter regions of interest of the brain | multiple visits up to 8 years post gene-therapy
  Measured to assess the pharmacodynamic activity of OTL-200 in neuronal metabolite ratio of NAA to Cr in white matter regions of interest of the brain post-treatment
Change from baseline in ARSA levels in total peripheral blood mononuclear cells (PBMCs) | 24 months and multiple visits up to 8 years post gene-therapy
  Measured to assess the pharmacodynamic activity of OTL-200 in circulating total PBMCs post-treatment
Change from baseline in ARSA levels in PB CD14+ | 24 months and multiple visits up to 8 years post gene-therapy
  Measured to assess the pharmacodynamic activity of OTL-200 in circulating CD14+ post-treatment
Change from baseline in ARSA levels in PB CD15+ | 24 months and multiple visits up to 8 years post gene-therapy
  Measured to assess the pharmacodynamic activity of OTL-200 in circulating CD15+ post-treatment
Neuronal metabolite ratios as compared to baseline, siblings and/or untreated historical controls (may include but not limited to Cho:Cr, mIns:Cr, Lac: Cr, Cho: NAA, NAA: H2O, Cho: H2O, mIns: H2O, Lac: H2O) in white matter regions of interest | 24 months and multiple visits up to 8 years post gene-therapy
  Measured to assess the pharmacodynamic activity of OTL-200 in neuronal metabolite ratios in white matter regions of interest of the brain post-treatment compared to siblings and/or untreated historical controls
Engraftment as measured by percent lentiviral positive (%LV+) in bone marrow (BM) progenitors | At D30 and multiple visits up to 8 years post gene-therapy
  Engraftment of transduced cells will be determined by measuring the percentage of hematopoietic colony-forming cells harboring the integrated vector by quantitative polymerase chain reaction (qPCR).
Vector copy number (VCN) in BM mononuclear cells | At D30 and multiple visits up to 8 years post gene-therapy
  Engraftment of transduced cells will be determined by measuring the VCN per genome in BM-derived cells.
VCN in Peripheral blood PBMCs | At D60 and multiple visits up to 8 years post gene-therapy
  Engraftment of transduced cells will be determined by measuring the VCN per genome in PBMCs.
Change in severity scale for brain magnetic resonance imaging (MRI) | 24 months and multiple visits up to 8 years post gene-therapy
  Brain MRI will be assessed using modified Loes Score and demyelination load on T1w, T2w and FLAIR imaging.
Change in neurocognitive function | 24 months and multiple visits up to 8 years post gene-therapy as compared to baseline
  Neurocognitive assessments will use Bayley Scale of Infant and Toddler Development (BSID), Wechsler Preschool and Primary Scale of Intelligence (WPPSI), Wechsler Intelligence Scale for Children (WISC), or Wechsler Adult Intelligence Scale (WAIS) according to the age of the participant to encompass performance, verbal, full scale IQ measures, processing speed and working memory indices
Change in full neurological clinical examination (NCE) | 24 months and multiple visits up to 8 years post gene-therapy
  Neurological examinations will be performed to evaluate the effect of OTL-200 on the onset or progression of MLD disease.
Change in Gross Motor Function Classification (GMFC)-MLD | 24 months and multiple visits up to 8 years post gene-therapy
  GMFC-MLD will evaluate the change in motor function according to seven clinically relevant levels of walking, sitting, locomotion, trunk and head control. The scoring range is from 0 (walking without support with quality of performance normal for age) to 6 (loss of any locomotion as well as loss of any head and trunk control).
Change in NCV | 24 months and multiple visits up to 8 years post gene-therapy
  NCV will be assessed by electroneurography which is a technique used to test and quantify the nerve conduction and impulse propagation along motor and sensory peripheral nerves.
Vineland Adaptive Behavior Scale (VABS) | 24 months and multiple visits up to 8 years post gene-therapy
  VABS will assess the individual's ability to undertake daily activities appropriate for their age group.
Conditioning regimen related toxicity and AEs | up to 8 years post gene-therapy
  To evaluate the safety and tolerability of the HSPC GT procedure.
Non-conditioning related AEs | up to 8 years post gene-therapy
  To evaluate the safety and tolerability of OTL-200.
Hematological reconstitution | By Day 60 post-gene therapy
  Hematological reconstitution defined as absolute neutrophil count [ANC] ≥ 500/µL and platelet count ≥20,000 platelets/μL with associated evidence of BM recovery
Incidence of infusion related reactions | up to 8 years post gene-therapy
  To evaluate the safety and tolerability of the HSPC GT procedure.
Immune response (e.g. anti-ARSA antibodies) | up to 8 years post gene-therapy
  Plasma samples will be collected for anti-ARSA antibody analysis
Abnormal Clonal Proliferation (ACP) | up to 8 years post gene-therapy
  Malignancy or ACP due to insertional oncogenesis will be evaluated using different tests and procedures.
Replication Competent Lentivirus (RCL | baseline, 1, 3, 6, and 12 months, then once a year up to 8 years post gene-therapy
  Molecular monitoring of RCL will be assessed via enzyme-linked immunosorbent assay (ELISA) test for serum human immunodeficiency virus (HIV) p24 antigen. A positive HIV p24 test result is subject to second level testing including: a) DNA PCR for vesicular stomatitis virus G (VSV-G) envelope (PBMC), and b) reverse transcription (RT)-PCR for serum HIV-pol ribonucleic acid (RNA) (plasma).
Integration Site analysis findings | 6, 12 months, then once a year up to 8 years post gene-therapy
  Detailed analysis of LV integrations will be performed on PB and BM cells, to monitor the nature and distribution of Integration Sites

CONTACTS AND LOCATIONS:
Overall Officials: Orchard Clinical Trials, Study Director — Orchard Therapeutics
Locations (1):
- Ospedale San Raffaele - Telethon Institute for Gene Therapy (OSR-TIGET), Milan, Italy